CLINICAL TRIAL: NCT03402932
Title: The Impact of Test Administration Method on Cognitive Screening Results in Older Individuals With Hearing Loss
Brief Title: Administration Method of Cognitive Screening in Older Individuals With Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jing Shen, Research Assistant Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 2R01DC012289 (NIH)
Record Dates: First submitted 2018-01-04; First posted 2018-01-18 (Actual); Results first posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Hearing Loss, Sensorineural; Cognitive Impairment
MeSH Terms: conditions — Hearing Loss, Sensorineural; Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Auditory Amplified-Visual (Experimental): This arm is designed to test the contrast between auditory amplified and visual conditions.
  Interventions: Other: Auditory amplified; Other: Visual
- Auditory Amplified-Unamplified (Experimental): This arm is designed to test the contrast between auditory amplified and unamplified conditions.
  Interventions: Other: Auditory amplified; Other: Auditory unamplified
- Auditory Unamplified-Visual (Experimental): This arm is designed to test the contrast between auditory unamplified and visual conditions.
  Interventions: Other: Visual; Other: Auditory unamplified
- Younger control group (Other): This arm is designed to validate the visual version by comparing to the auditory version in a group of younger normal hearing controls.
  Interventions: Other: Visual; Other: Auditory unamplified

INTERVENTIONS:
Other: Auditory amplified — The cognitive test will be administered using a computer-based signal processing to amplify the instruction. The presentation level is customized to the individual's hearing thresholds.
  Arms: Auditory Amplified-Unamplified; Auditory Amplified-Visual
Other: Visual — The cognitive test will be administered visually by using timed computer slides.
  Arms: Auditory Amplified-Visual; Auditory Unamplified-Visual; Younger control group
Other: Auditory unamplified — The cognitive test will be administered by using a generic presentation level that simulates a normal conversational level.
  Arms: Auditory Amplified-Unamplified; Auditory Unamplified-Visual; Younger control group

SUMMARY:
The objectives of the current project aim to determine whether a more controlled amplification method or a visual administration has an effect on hearing impaired older individuals' cognitive test scores.

DETAILED DESCRIPTION:
Aim 1 is to create a visually administered condition of a cognitive test and to validate this condition in comparison to the auditory administration. Data will be collected from younger individuals with normal hearing. Each younger individual is tested using both visual and auditory condition and the scores are compared across the two conditions. It is anticipated that the scores will not be significantly different between the two conditions.

Aim 2 is to examine the test condition effect on cognitive testing results in older individuals with hearing loss. The three test conditions include auditory unamplified, auditory amplified, and visual. Each older individual will be tested using two different test conditions. It is predicted the auditory amplified and visual administrations will alleviate the cognitive load associated with hearing difficulty and lead to improved performance on the test.

ELIGIBILITY:
Inclusion Criteria:

* Have sensorineural hearing loss
* Have normal or corrected-to-normal vision

Exclusion Criteria:

* Have conductive hearing loss;
* Have history of otologic or neurologic disorders
* Have dementia
* Non-native speakers of English

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hearing Aid Laboratory, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
The results will be shared in the form of presentations and publications. Study protocol is available upon request.

REFERENCES:
- [Background] Jorgensen LE, Palmer CV, Pratt S, Erickson KI, Moncrieff D. The Effect of Decreased Audibility on MMSE Performance: A Measure Commonly Used for Diagnosing Dementia. J Am Acad Audiol. 2016 Apr;27(4):311-23. doi: 10.3766/jaaa.15006. PMID 27115241
- [Background] Guerreiro MJS, Van Gerven PWM. Disregarding hearing loss leads to overestimation of age-related cognitive decline. Neurobiol Aging. 2017 Aug;56:180-189. doi: 10.1016/j.neurobiolaging.2017.05.001. Epub 2017 May 10. PMID 28559106
- [Background] Lin FR, Yaffe K, Xia J, Xue QL, Harris TB, Purchase-Helzner E, Satterfield S, Ayonayon HN, Ferrucci L, Simonsick EM; Health ABC Study Group. Hearing loss and cognitive decline in older adults. JAMA Intern Med. 2013 Feb 25;173(4):293-9. doi: 10.1001/jamainternmed.2013.1868. PMID 23337978
- [Background] Dupuis K, Pichora-Fuller MK, Chasteen AL, Marchuk V, Singh G, Smith SL. Effects of hearing and vision impairments on the Montreal Cognitive Assessment. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2015;22(4):413-37. doi: 10.1080/13825585.2014.968084. Epub 2014 Oct 17. PMID 25325767

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant event after andnrollment, prior to assignment
Groups:
- Group1: Auditory -Visual (Younger Adults w/ Normal Hearing): A group of younger adults with normal hearing is included to validate the visual version of the tests
- Group2: Amplified-Visual (Older Adults w/ Hearing Loss): Auditory amplified: The cognitive test was administered using a computer-based signal processing to amplify the instruction. The presentation level was customized to the individual's hearing thresholds.
  Visual: The cognitive test was administered visually by using timed computer slides.
- Group3: Amplified-Unamplified (Older Adults w/ Hearing Loss): Auditory amplified: The cognitive test was administered using a computer-based signal processing to amplify the instruction. The presentation level was customized to the individual's hearing thresholds.
  Auditory unamplified: The cognitive test was administered by using a generic presentation level that simulates a normal conversational level.
- Group4: Visual-Unamplified (Older Adults w/ Hearing Loss): Visual: The cognitive test was administered visually by using timed computer slides.
  Auditory unamplified: The cognitive test was administered by using a generic presentation level that simulates a normal conversational level.
Period: Overall Study
Arm/Group | Group1: Auditory -Visual (Younger Adults w/ Normal Hearing) | Group2: Amplified-Visual (Older Adults w/ Hearing Loss) | Group3: Amplified-Unamplified (Older Adults w/ Hearing Loss) | Group4: Visual-Unamplified (Older Adults w/ Hearing Loss)
Started | 13 | 8 | 8 | 8
Completed | 13 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group1: Younger Control (Auditory Unamplified - Visual): This arm is for validating the visual version of the tests with younger individuals with normal hearing.
  Visual: The cognitive test was administered visually by using timed computer slides.
  Auditory unamplified: The cognitive test was administered by using a generic presentation level that simulates a normal conversational level.
- Group2: Auditory Amplified - Visual: Auditory amplified: The cognitive test was administered using a computer-based signal processing to amplify the instruction. The presentation level was customized to the individual's hearing thresholds.
  Visual: The cognitive test was administered visually by using timed computer slides.
- Group3: Auditory Amplified - Unamplified: Auditory amplified: The cognitive test was administered using a computer-based signal processing to amplify the instruction. The presentation level was customized to the individual's hearing thresholds.
  Auditory unamplified: The cognitive test was administered by using a generic presentation level that simulates a normal conversational level.
- Group4: Auditory Unamplified - Visual: Visual: The cognitive test was administered visually by using timed computer slides.
  Auditory unamplified: The cognitive test was administered by using a generic presentation level that simulates a normal conversational level.
- Total: Total of all reporting groups
Arm/Group | Group1: Younger Control (Auditory Unamplified - Visual) | Group2: Auditory Amplified - Visual | Group3: Auditory Amplified - Unamplified | Group4: Auditory Unamplified - Visual | Total
Number analyzed (Participants) | 13 | 8 | 8 | 8 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 0 | 0 | 0 | 13
  >=65 years | 0 | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.69 (2.78) | 77 (5.91) | 73.37 (4.12) | 73.75 (6.35) | 28.5 (1.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 5 | 5 | 24
  Male | 3 | 4 | 3 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 12 | 8 | 8 | 8 | 36
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 8 | 8 | 8 | 36

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Screening Results (Montreal Cognitive Assessment)
Description: The cognitive screening test of Montreal Cognitive Assessment (MoCA) was administered to 4 groups with different administration method conditions (see arms/groups table).
  MoCA is s standardized cognitive screening tool for mild cognitive impairment and dementia. The total score was used as outcome measure of this study and this score ranges from 0-30, with higher score being better performance.
Time Frame: The outcome measure was assessed immediately after the test. This applies to both conditions for all the arms.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group1: Auditory Unamplified -Visual (Younger Adults): Younger adults with normal hearing group was included to validate the visual version of the test.
  The auditory administration was unamplified. The visual administration had all test material visually presented.
- Group2: Amplified-Visual (Older Adults w/ Hearing Loss): Auditory amplified: The cognitive test was administered using a computer-based signal processing to amplify the instruction. The presentation level was customized to the individual's hearing thresholds.
  Visual administration presented all test material visually.
- Group3: Amplified-Unamplified (Older Adults w/ Hearing Loss): Auditory amplified: The cognitive test was administered by using customized amplification.
  Auditory unamplified: The cognitive test was administered by using a generic presentation level that simulates a normal conversational level.
Arm/Group | Group1: Auditory Unamplified -Visual (Younger Adults) | Group2: Amplified-Visual (Older Adults w/ Hearing Loss) | Group3: Amplified-Unamplified (Older Adults w/ Hearing Loss) | Group4: Visual-Unamplified (Older Adults w/ Hearing Loss)
Number analyzed (Participants) | 13 | 8 | 8 | 8
score on a scale
  Condition 1 | 28.69 (1.2) | 22.37 (2.82) | 23.375 (2.34) | 23 (2.82)
  Condition 2 | 28.30 (1.13) | 23.5 (2.91) | 24.125 (1.26) | 22.12 (2.8)

2. Secondary Outcome: Auditory Working Memory Performance
Description: Older individuals were presented with lists of words and instructed to repeat them back. After each word list, they had to recall the words.
Time Frame: The outcome measure will be assessed immediately after the test.
Measure: Mean (Standard Deviation); unit: percentage of correct recall
Arm/Group | Group1: Younger Control (Auditory Unamplified - Visual) | Group2: Auditory Amplified - Visual | Group3: Auditory Amplified - Unamplified | Group4: Auditory Unamplified - Visual
Number analyzed (Participants) | 13 | 8 | 8 | 8
percentage of correct recall
  Condition 1 | 82.88 (6.7) | 72.3 (7.1) | 69.1 (8.2) | 57.5 (11.5)
  Condition 2 | 82.11 (7.6) | 66.9 (9.66) | 64.5 (11.4) | 61.3 (14.5)

ADVERSE EVENTS:
Time Frame: The outcome measures are behavioral measures (e.g., cognitive screening test scores) and were collected within a short period of time (2 hours).
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- Group1: Younger Auditory Unamplified - Visual; Group2: Auditory Amplified - Visual; Group3: Auditory Amplified - Unamplified; Group4: Auditory Unamplified - Visual: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Group1: Younger Auditory Unamplified - Visual | Group2: Auditory Amplified - Visual | Group3: Auditory Amplified - Unamplified | Group4: Auditory Unamplified - Visual
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT03402932/SAP_000.pdf
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT03402932/Prot_001.pdf